CLINICAL TRIAL: NCT06250751
Title: Behavioral Exercise TRaining for Medically Underserved Men Undergoing Androgen Deprivation Therapy for Prostate Cancer (BETR-PC)
Brief Title: Behavioral Exercise TRaining for Men Undergoing Androgen Depr Therapy for Prostate Ca
Acronym: BETR-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23-20769; HM20028651 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Exercise; Prostate Cancer; Androgen Deprivation Therapy (ADT); Home Based Exercise Intervention
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — DNER protein, human; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral exercise training (BET) to introduce behavioral skills for adopting an exercise program (Experimental): Single-arm, ORBIT-prospective, multicenter, nonblinded clinical trial, feasibility pilot. The BET intervention will be delivered and refined over 12 weeks. The protocol aim is to enroll men from the same representative groups of underserved men in groups of 5-10, to foster social support and group cohesion.
  Interventions: Behavioral: Behavioral Exercise Training (BET) intervention

INTERVENTIONS:
Behavioral: Behavioral Exercise Training (BET) intervention — Introduce and refine concept of exercise and cardiovascular health by initiating walking or cycling and provide behavioral counseling sessions to foster support for adoption and maintenance of exercise, and to troubleshoot barriers. During the first two weeks, the study team will meet with participants twice per week (virtually) to introduce the intervention, familiarize men with the exercise program, exercise logs, resistance bands for strength training. Contact will drop to once per week during weeks 3-8 (total=10 contacts in weeks 1-8). Behavioral counseling will be delivered by the PI or the study coordinator for 30-40 minutes prior to 20-30 mins of an individual or group-based strength training class.

SUMMARY:
To refine a remote behavioral exercise training intervention for testing in a larger randomized trial.

DETAILED DESCRIPTION:
Determine feasibility of recruiting a sample of medically underserved prostate cancer patients undergoing treatment with Androgen Deprivation Therapy (ADT) to a remotely delivered (i.e., home-based) exercise intervention and determine the interventions acceptability.

ELIGIBILITY:
Inclusion Criteria:

To be eligible men, transwomen or non-binary individuals must meet the following criteria:

* Be diagnosed with stage II/III/IV prostate cancer
* Be currently undergoing treatment with ADT (intermittent or prolonged)
* Have completed local curative-intent treatment, including prostatectomy or definitive radiation
* Be >40 years of age if non-Hispanic Black or rural dwelling; Otherwise >60 years of age up to 85
* Be willing to give an informed consent and sign a HIPAA authorization form
* Not have any hearing or sight impairments that result in the inability to use the telephone or hear normal conversation
* Must be able to join an intervention group by personal computer, smartphone or telephone call and should agree to recording of an interview
* Be without any serious medical condition that precludes safe participation in an exercise program
* Speak English.
* Meet protocol definition of medically underserved: which is consider medically underserved patients to be a) older men (>75 years), b) men who live in rural zip code areas, or c) men who identify as being non-Hispanic Black. They may also be at the intersectionality of these groups (i.e., older Black men living in a rural zip code area).

Ages: 41 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of trial by assessing the recruitment rate | Day 1
  The number of participants that enroll
Feasibility of trial by assessing the retention rate | 12 Weeks
  The number of participants that complete greater than 80% of the planned assessments
Acceptability of the trial by assessing the retention rate | 12 Weeks
  Number of participants that adhere to and complete the intervention

SECONDARY OUTCOMES:
Physical activity levels using accelerometry (ActivPAL, Actigraph) | Baseline, 8 Weeks, and 12 Weeks
  An ActivPAL is a small, previously validated thigh-worn device that continuously measures physical activity, sitting time or movement. An Actigraph is a small wrist worn device that continuously measures physical activity intensity (i.e., exercise intensity), sleep time or movement.
Physical activity levels using the Godin-Leisure Time Exercise Questionnaire (GLTEQ). | Baseline, 8 Weeks, and 12 Weeks
  The average of the scores for participants using the GLTEQ is a 3-item measure used to classify participant's activity levels per week. The Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light). The Godin scale score = 24 units or more=active, 14-23 units= moderately active, and less than 14 unites = insufficiently active/ sedentary.
Submaximal exercise capacity assessed with the 6-minute walk test. | Baseline, 8 Weeks, and 12 Weeks
  Measuring changes in a 6 minute walk distance. The participant has a goal to walk as fast, but safely, as possible without running for a period of 6 minutes.
Physical function as assessed with the short physical performance battery (SPPB). | Baseline, 8 Weeks, and 12 Weeks
  Short Physical Performance Battery (Short Physical Performance Battery (SPPB) is a battery of 3 tests (standing balance, gait speed and char stands) that are combined to assess overall physical function. Each test is scored on a scale of 1-4 with 4 being reflective of good function and 0 of poor function. Overall scores of 10 or less are reflective of mobility limitations.
Lower body strength assessed with a 30 seconds chair stand test. | Baseline, 8 Weeks, and 12 Weeks
  Participants will be first asked to stand from a sitting position without using their arms. If they can perform the task, they will then be asked to stand up and sit down as many times as possible in a 30 second period. The greater the number of chair stands the better the lower body strength.
Upper body strength assessed with a grip strength dynamometer. | Baseline, 8 Weeks, and 12 Weeks
  Grip strength will be assessed using an isometric handgrip dynamometer while the participant is seated with the head facing straight ahead. The elbow should be bent at a 90-degree angle and the wrist should be at the mid-prone position. The participant should exert maximally and quickly (about 1 second) and two trials should be made alternately with each hand, with at least 30 seconds between trials for the same hand (recorded in kilograms).
Self-efficacy for exercise using the exercise self-efficacy scale (EXSE) to assess socioecological model constructs as multilevel factors associated with physical activity levels and behavioral patterns | Baseline, 8 Weeks, and 12 Weeks
  The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future. For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Social support for exercise scale to assess socioecological model constructs as multilevel factors associated with physical activity levels and behavioral patterns | Baseline, 8 Weeks, and 12 Weeks
  Assessment of the level of support individuals making health-behavior changes (exercise) felt they were receiving from family and friends.
  Family Participation: sum items 11 - 16 and 20 - 23 Family Rewards and Punishment (an optional scale): sum items 17 - 19 Friend Participation: sum items 11 - 16 and 20 - 23
  Higher scores reflect more support.
Walk Score to assess socioecological model constructs as multilevel factors associated with physical activity levels and behavioral patterns | Baseline, 8 Weeks, and 12 Weeks
  Walk Score measures the walkability of any address using a patented system. For each address, Walk Score analyzes hundreds of walking routes to nearby amenities. Points are awarded based on the distance to amenities in each category. Amenities within a 5 minute walk (.25 miles) are given maximum points.
  90-100 is a good walk score 70-89 is very walkable 50-69 is somewhat walkable 0-49 is car dependent
Assess health-related quality of life (HRQL) using the Functional Assessment of Cancer Therapy-Fatigue scale (FACIT-fatigue) | Baseline, 8 Weeks, and 12 Weeks
  The FACIT-fatigue scale is a 13-item scale that has been widely used in many studies to assess cancer related fatigue
  Scores range from 0-52 with higher scores indicating better quality of life.
Assess disease specific quality of life (HRQL) using the 42-item Functional Assessment of Cancer Treatment-Prostate (FACT-P) | Baseline, 8 Weeks, and 12 Weeks
  The FACT-P measure is composed of the FACT-General which assesses four primary HRQOL domains: physical well-being , functional well-being, social well-being, and emotional well-being and an additional component for prostate specific concerns.
  Scores range from 0-156 with higher scores reflecting better quality of life
Assess health-related quality of life (HRQL) using the the MOS 36-item Short Form Health Survey (SF-36) | Baseline, 8 Weeks, and 12 Weeks
  The SF-36 is perhaps the most widely used measure of health status and includes domains of vitality and physical function.
  The SF-36 has 8 subdomains (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health). Each scale item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively with 100 higher quality of life.
Assess health-related quality of life (HRQL) using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue Scale 4a | Baseline, 8 Weeks, and 12 Weeks
  PROMIS - Fatigue is a validated self-report measure of fatigue among patients diagnosed with cancer and higher scores indicate a lower level of fatigue. All scores are on a T-score distribution with a mean of 50 and standard deviation of 10.
Assess health-related quality of life (HRQL) using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function Scale 4a | Baseline, 8 Weeks, and 12 Weeks
  PROMIS - Physical function is a validated self-report measure of physical function among patients diagnosed with cancer and higher scores indicate better functioning. All scores are on a T-score distribution with a mean of 50 and standard deviation of 10.
Assess health-related quality of life (HRQL) using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety Scale 4a | Baseline, 8 Weeks, and 12 Weeks
  PROMIS - Anxiety is a validated self-report measure of physical function among patients diagnosed with cancer and higher scores indicate better functioning. All scores are on a T-score distribution with a mean of 50 and standard deviation of 10.
Assess health-related quality of life (HRQL) using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression Scale 4a | Baseline, 8 Weeks, and 12 Weeks
  PROMIS - Depression is a validated self-report measure of physical function among patients diagnosed with cancer and higher scores indicate better functioning. All scores are on a T-score distribution with a mean of 50 and standard deviation of 10.
Assess health-related quality of life (HRQL) using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Scale 4a | Baseline, 8 Weeks, and 12 Weeks
  PROMIS - Sleep disturbance is a validated self-report measure of physical function among patients diagnosed with cancer and higher scores indicate better functioning. All scores are on a T-score distribution with a mean of 50 and standard deviation of 10.
Assess health-related quality of life (HRQL) using Social Determinants of Health | Baseline, 8 Weeks, and 12 Weeks
  Social Determinants of Health (SDOH) questionnaire is a self-administered questionnaire used to examine education and income variables in relation to cardiovascular risk. The questionnaire is administered at the baseline visit. We will also ask about difficult paying for basics and experience of racial discrimination at 3- and 6-month follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lucas, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No